CLINICAL TRIAL: NCT02925338
Title: OBSERVATOIRE NATIONAL D'UTILISATION D'INFLECTRA™ EN VIE RÉELLE.
Brief Title: National Observational Study On The Use Of Inflectra™ An Infliximab Biosimilar In Real Life
Acronym: ReFLECT
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C1231004; REFLECT (Other: Alias Study Number)
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Results first posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Crohn Disease; Ulcerative Colitis; Rheumatoid Arthritis; Ankylosing Spondylitis; Psoriatic Arthritis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients treated with Inflectra
  Interventions: Other: QOL questionaire

INTERVENTIONS:
Other: QOL questionaire — Health assessment questionnaire disability index for rheumatoid polyarthritis questionnaire

SUMMARY:
National, prospective, multicentre observational study designed for eligible patients treated with Inflectra.

Its objectives are to describe under real conditions of use, the profile of patients treated with Inflectra and the response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients treated with Inflectra™ regardless of treatment phase in one of the following indications consistent with the SPC: Crohn's Disease, ulcerative colitis, rheumatoid arthritis, ankylosing spondylitis or psoriatic arthritis.
* Paediatric patients (children and adolescents between 6 and 17 years old) treated with Inflectra™, regardless of treatment phase from the time when Inflectra™ is prescribed in accordance with the indications listed in the SPC Crohn's Disease or ulcerative colitis Patients (or their legal representatives) who have received information (verbally and in writing) about the study and agreed to take part in it.
* Patients who have given their agreement for their clinical data and their medical file to be accessed by signing the information leaflet.

Exclusion Criteria:

* Patients who refuse access to their medical file for collection of: their medical data
* Patients not treated with Inflectra™.
* Patients treated with Inflectra™ for psoriasis.
* Patients with a past history of hypersensitivity to infliximab, to other murine proteins or to one of the excipients in Inflectra™.
* Patients with tuberculosis or any other severe infection such as sepsis, abscess or opportunistic infection .
* Patients with moderate to severe heart failure (NYHA III/IV)

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients treated with Inflectra™ regardless of treatment phase in one of the following indications consistent with the SPC: Crohn's Disease, ulcerative colitis, rheumatoid arthritis, ankylosing spondylitis or psoriatic arthritis.
  Paediatric patients (children and adolescents between 6 and 17 years old) treated with Inflectra™, regardless of treatment phase from the time when Inflectra™ is prescribed in accordance with the indications listed in the SPC Crohn's Disease or ulcerative colitis
Sampling Method: Probability Sample
Enrollment: 1431 (Actual)
Dates: Start 2016-10-19 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (67):
- France (67):
  - Hopitaux Universitaires de Strasbourg - Hopital de Hautepierre, Strasbourg, Alsace
  - Service de rhumatologie - CHU Nantes, Hopital Hotel Dieu, Nantes, Loire-atlantique
  - Centre Hospitalier Universitaire Gabriel Montpied, Clermont-Ferrand, Puy-de-dôme
  - Centre Hospitalier du Pays d'Aix, Aix-en-Provence
  - Chi Aix Pertuis, Aix-en-Provence
  - Centre Hospitalier de la Cote Basque, Bayonne
  - Centre Hospitalier Regional de Besancon, Service de Gastrologie, Besançon
  - CHU Jean Minjoz, Besançon
  - Hopital Saint Andre - Chu Bordeaux, Bordeaux
  - Centre Hospitalier Universitaire de Bordeaux - Hopital Pellegrin, Bordeaux
  - CHU - Hôpital Pellegrin-tripode, Bordeaux
  - Clinique Jean Vila, Bruges
  - Clinique Jean Vilar, Bruges
  - Centre Hospitalier Universitaire (CHU) de Caen - Hopital Cote de Nacre, Caen
  - Centre Hospitalier de Cannes Hopital Pierre Nouveau, Cannes
  - Centre Hospitalier de Cannes, Cannes
  - Ch de Cannes Hopital Pierre Nouveau, Cannes
  - Centre Hospitalier Carcassonne, Service de Rhumatologie, Carcassonne
  - Centre Hospitalier de Cholet Service d'Hépato-Gastro-Entérologie, Cholet
  - Centre Hospitalier de Cholet, Cholet
  - Centre Hospitalier Estaing, Service de Medicine Interne, Clermont-Ferrand
  - Hopital Beaujon, Clichy
  - Centre Hospitalier, Contamine Sur Avre
  - Chu Henri Mondor, Créteil
  - CHU de Grenoble - Hopital Sud, Échirolles
  - Hopital Nord, Grenoble
  - CHU De Grenoble, Grenoble
  - CHD Vendee, La Roche-sur-Yon
  - Centre Hospitalier Universitaire Grenoble Alpes, La Tronche
  - CHU Grenoble Alpes, La Tronche
  - Centre Hospitalier de Lille Hopital Roger Salengro, Lille
  - CHU Limoges - Hôpital Dupuytren, Limoges
  - Hospital Huriez, CHRU de Lille, Little Cedex
  - Hopital Saint Philibert, Lomme
  - Hopital Edouard Herriot Pav H, Lyon
  - Centre Hospitalier, Metz-Tessy
  - CHG Montauban, Montauban
  - Groupe Hospitalier du Havre, Montivilliers
  - Centre Hospitalier de Montpellier Hopital Saint Eloi, Montpellier
  - CHU de Montpellier - Saint Eloi, Montpellier
  - CHU de MONTPELLIER HOPITAL LAPEYRONIE, Montpellier
  - CHU, Montpellier
  - CHU Nice-Hopital Archet I, Nice
  - Hopital de l'Archet, Nice
  - CHU Nimes, Nîmes
  - Hopital Cochin, Paris
  - Hôpital Cochin, Paris
  - Hopital Claude Bichat, Paris
  - Hôpital Haut-Lévêque, Pessac
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Hopital Lyon Sud, Pierre-Bénite
  - Hopital Robert Debre, Service d'Hepato-gastro-enterologie et de Cancerologie Digestive, Reims
  - Hopital Robert Debre, Service D'Hepato-gastro-enterolo, Reims
  - CHU de Rouen, Rouen
  - CHRU Charles Nicolle, Rouen
  - Service Rhumatologie, Saint-Etienne
  - Centre Hospitalier Universitaire (CHU) de Saint-Etienne - Hopital Nord, Saint-Priest-en-Jarez
  - Hopital Nord, Saint-Priest-en-Jarez
  - Fondation Maison Sante Bagatelle, Gastro Enterologie, Talence
  - Centre Hospitalier de la Gespe, Tarbes
  - Hopital du Leman, Thonon-les-Bains
  - Hopitaux du Leman, Thonon-les-Bains
  - Hopital Purpan, Toulouse
  - Hopital Rangueil, Toulouse
  - Hopital des Hauts Clos, Troyes
  - Chu Brabois, Vandœuvre-lès-Nancy
  - Hopital Saint Nicolas, Vitré

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Marotte H, Cantagrel A, Coury F, Schaeverbeke T, Assing M, Kessouri M, Brault Y, Fautrel B. Real-World Effectiveness and Safety of Infliximab Biosimilar CT-P13 for Rheumatic Diseases: A National Observational Cohort Study (ReFLECT). Adv Ther. 2025 Sep;42(9):4659-4680. doi: 10.1007/s12325-025-03304-6. Epub 2025 Jul 28. PMID 40720061
- [Derived] Laharie D, Bouhnik Y, Vuitton L, Biron A, Pierron G, Brault Y, Assing M, Bouzidi A, Amiot A, Nancey S. Real-world effectiveness and safety of CT-P13, an infliximab biosimilar, for inflammatory bowel diseases: A prospective national observational cohort study (ReFLECT study). Clin Res Hepatol Gastroenterol. 2024 Dec;48(10):102483. doi: 10.1016/j.clinre.2024.102483. Epub 2024 Oct 22. PMID 39448029
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1231004

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who were being treated with Inflectra or who initiated Inflectra or switched from infliximab reference to Inflectra in real world practice for following indications, in conformity to summary of product characteristics (SmPC): adult participants with crohn's disease (CD), ulcerative colitis (UC), rheumatoid arthritis (RA), ankylosing spondylitis (SpA) or psoriatic arthritis (PA); pediatric participants with CD or UC, were observed for 2 years post inclusion in this study.
Pre-assignment Details: Total 1431 participants were enrolled in this study, however only 1426 participants received the treatment. 5 participants did not receive the treatment due to major protocol deviations.
Groups:
- Crohn's Disease (CD): Adult participants diagnosed with moderately to fistulizing active CD received 5 milligrams per kilogram (mg/kg) of Inflectra as an intravenous (IV) infusion followed by additional 5 mg/kg infusion at 2 weeks (for moderate to severely active CD) and at 2 weeks and 6 weeks (for fistulizing active) after the first infusion. Participants who responded to the treatment received additional infusion of 5 mg/kg at 6 weeks after the initial dose, followed by infusions every 8 weeks or infusion of 5 mg/kg if signs and symptoms of the disease. Pediatric participants diagnosed with CD received 5 mg/kg given as an IV infusion followed by additional 5 mg/kg infusion doses at 2 and 6 weeks after the first infusion, then every 8 weeks thereafter. Participants were observed for 2 years in this study.
- Ulcerative Colitis (UC): Adult and pediatric participants included in this arm were diagnosed with UC and received 5 mg/kg of Inflectra as an IV infusion followed by additional 5 mg/kg infusion doses at 2 and 6 weeks after the first infusion, then every 8 weeks thereafter. Participants were observed for 2 years in this study.
- Rheumatoid Arthritis (RA): Adult participants included in this arm were diagnosed with RA and received 3 mg/kg of Inflectra as an IV infusion followed by additional 3 mg/kg infusion doses at 2 and 6 weeks after the first infusion, then every 8 weeks thereafter. Inflectra was administered in combination with methotrexate. Participants were observed for 2 years in this study.
- Ankylosing Spondylitis (SpA): Adult participants included in this arm were diagnosed with SpA and received 5 mg/kg of Inflectra as an IV infusion followed by additional 5 mg/kg infusion doses at 2 and 6 weeks after the first infusion, then every 6 to 8 weeks. Participants were observed for 2 years in this study.
- Psoriatic Arthritis (PA): Adult participants included in this arm were diagnosed with PA and received 5 mg/kg of Inflectra as an IV infusion followed by additional 5 mg/kg infusion doses at 2 and 6 weeks after the first infusion, then every 8 weeks thereafter. Participants were observed for 2 years in this study.
Period: Overall Study
Arm/Group | Crohn's Disease (CD) | Ulcerative Colitis (UC) | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
Started | 547 | 230 | 142 | 411 | 96
Adult Population | 530 | 221 | 142 | 411 | 96
Pediatric Population | 17 | 9 | 0 | 0 | 0
Completed | 321 | 119 | 78 | 251 | 66
Not Completed | 226 | 111 | 64 | 160 | 30
Not completed — Death | 0 | 2 | 1 | 0 | 0
Not completed — Lost to Follow-up | 30 | 10 | 1 | 16 | 3
Not completed — Withdrawal by Subject | 3 | 0 | 3 | 2 | 2
Not completed — Missing | 38 | 27 | 0 | 3 | 2
Not completed — Participant's Decision | 11 | 7 | 3 | 8 | 1
Not completed — Treatment Discontinuation | 144 | 65 | 56 | 131 | 22

BASELINE CHARACTERISTICS:
Population: Analysis population included all enrolled participants treated with Inflectra.
Groups:
- Crohn's Disease (CD): Adult participants diagnosed with moderately to fistulizing active CD received 5 mg/kg of Inflectra as an IV infusion followed by additional 5 mg/kg infusion at 2 weeks (for moderate to severely active CD) and at 2 weeks and 6 weeks (for fistulizing active) after the first infusion. Participants who responded to the treatment received additional infusion of 5 mg/kg at 6 weeks after the initial dose, followed by infusions every 8 weeks or infusion of 5 mg/kg if signs and symptoms of the disease. Pediatric participants diagnosed with CD received 5 mg/kg given as an IV infusion followed by additional 5 mg/kg infusion doses at 2 and 6 weeks after the first infusion, then every 8 weeks thereafter. Participants were observed for 2 years in this study.
- Total: Total of all reporting groups
Arm/Group | Crohn's Disease (CD) | Ulcerative Colitis (UC) | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA) | Total
Number analyzed (Participants) | 547 | 230 | 142 | 411 | 96 | 1426
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.4 (14.2) | 42.3 (17.9) | 61.5 (10.9) | 48.1 (13.1) | 53.4 (14.1) | 44.8 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 281 | 103 | 107 | 169 | 56 | 716
  Male | 266 | 127 | 35 | 242 | 40 | 710
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] — BMI of participants in kilogram (kg)/square meter (m^2) was reported for this baseline measure. Population: Here, "Overall Number of Participants Analyzed" signifies participants analyzed for this baseline measure.
  Kg/m^2
    number analyzed (Participants) | 541 | 224 | 132 | 393 | 95 | 1385
    (all) | 24.01 (5.52) | 24.29 (4.72) | 27.12 (5.68) | 26.52 (5.44) | 29.26 (6.71) | 25.42 (5.71)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Without Treatment Failure During 2-Years of Observation
Description: Treatment failure was defined as permanent discontinuation of the Inflectra treatment due to intolerance and/or permanent discontinuation of treatment due to absence of response according to the physician's assessment, or death of the participant related to Inflectra. In this outcome measure percentage of participants without treatment failure and whose data were missing are reported.
Time Frame: 2 years post inclusion in the study
Population: Analysis population included all enrolled participants treated with Inflectra.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Crohn's Disease (CD) | Ulcerative Colitis (UC) | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
Number analyzed (Participants) | 547 | 230 | 142 | 411 | 96
Percentage of participants
  Without Treatment Failure | 59.2 [55.1 to 63.4] | 53.5 [47.0 to 59.9] | 53.5 [45.3 to 61.7] | 61.1 [56.4 to 65.8] | 64.6 [55.0 to 74.2]
  Missing Data | 19.2 [15.9 to 22.5] | 21.3 [16.0 to 26.6] | 7.7 [3.3 to 12.1] | 14.4 [11.0 to 17.7] | 9.4 [3.5 to 15.2]

2. Primary Outcome: Number of Participants With Pre-treatment Assessment Prior to Initiation of Inflectra Treatment (Anti-Tumor Necrosis Factor [TNF] Aplha) Therapy
Description: Pre-treatment assessment was a check-list with the set of measures determined by the physician to check the eligibility of a participant before initiation of treatment. Physician recorded as "Yes" if a participant was eligible for initiation of treatment and "No" if a participant was not eligible to initiate a treatment. In this outcome measure, number of participants whose pre-treatment assessment were performed prior to initiation of Inflectra are reported and whose data were missing are reported.
Time Frame: Data collected and recorded at study inclusion visit
Population: Analysis population included all enrolled participants treated with Inflectra.
Measure: Count of Participants; unit: Participants
Arm/Group | Crohn's Disease (CD) | Ulcerative Colitis (UC) | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
Number analyzed (Participants) | 547 | 230 | 142 | 411 | 96
Participants
  Had Pre-treatment Assessment | 458 | 177 | 118 | 355 | 86
  Missing Data | 5 | 4 | 2 | 2 | 0

3. Primary Outcome: Time Between Diagnosis and Inclusion in Study
Time Frame: Data collected and recorded at study inclusion visit
Population: Analysis population included all enrolled participants treated with Inflectra. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure with non-missing data.
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Crohn's Disease (CD) | Ulcerative Colitis (UC) | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
Number analyzed (Participants) | 546 | 230 | 142 | 407 | 95
Years | 10.05 (9.51) | 8.77 (8.56) | 15.18 (10.13) | 13.58 (10.26) | 11.50 (8.42)

4. Primary Outcome: Time Between Diagnosis and the First Inflectra Infusion
Time Frame: Data collected and recorded at study inclusion visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Crohn's Disease (CD) | Ulcerative Colitis (UC) | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
Number analyzed (Participants) | 535 | 224 | 142 | 402 | 93
Years | 9.37 (9.67) | 8.22 (8.66) | 14.39 (10.11) | 12.80 (10.29) | 10.78 (8.42)

5. Primary Outcome: Number of Participants Who Received Biotherapy Other Than Inflectra Before Inclusion in the Study
Description: Type of biotherapies received by participants before inclusion in the study were: anti-TNF alpha (remicade/ adalimumab/ golimumab / etanercept/ rituximab); anti-integrin (vedolizumab); immunosuppressant (abatacept); interleukin inhibitor (anakinra / tocilizumab); anti interleukin (IL) 12 and anti IL-23 (ustekinumab); and other. In this outcome measure number of participants who received biotherapies other than Inflectra and whose data were missing are reported.
Time Frame: Data collected and recorded at study inclusion visit
Population: Analysis population included all enrolled participants treated with Inflectra.
Measure: Count of Participants; unit: Participants
Arm/Group | Crohn's Disease (CD) | Ulcerative Colitis (UC) | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
Number analyzed (Participants) | 547 | 230 | 142 | 411 | 96
Participants
  Received Biotherapy | 347 | 146 | 116 | 344 | 81
  Missing Data | 4 | 2 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Reasons for Discontinuation of Previous Biotherapy
Description: Type of previous biotherapies included were: anti-TNF alpha (infliximab/adalimumab/etanercept/golimumab), selective immuno-suppressant (vedolizumab/abatacept), interleukin inhibitor (anakinra/ustekinumab/tocilizumab), and other. In this outcome measure, number of participants who discontinued previous biotherapy are reported according to reason of discontinuations.
Time Frame: Data collected and recorded at study inclusion visit
Population: Analysis population included all enrolled participants treated with Inflectra. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Crohn's Disease (CD) | Ulcerative Colitis (UC) | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
Number analyzed (Participants) | 347 | 146 | 116 | 344 | 81
Participants
  Missing | 13 | 5 | 5 | 29 | 6
  Loss of Efficacy | 80 | 35 | 19 | 52 | 14
  Primary Non-response | 25 | 40 | 16 | 49 | 10
  Intolerance | 42 | 5 | 9 | 23 | 9
  Remission | 0 | 0 | 0 | 0 | 1
  Switch Inflectra | 164 | 52 | 57 | 166 | 32
  Other | 23 | 9 | 10 | 25 | 9

7. Primary Outcome: Duration of Previous Biotherapies
Description: Type of previous biotherapies included were: anti-TNF alpha (infliximab/adalimumab/etanercept/golimumab), selective immuno-suppressant (vedolizumab/abatacept), interleukin inhibitor (anakinra/ustekinumab/tocilizumab), and other.
Time Frame: Data collected and recorded at study inclusion visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Crohn's Disease (CD) | Ulcerative Colitis (UC) | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
Number analyzed (Participants) | 339 | 143 | 116 | 338 | 79
Months | 51.3 (43.1) | 33.2 (38.2) | 81.0 (55.8) | 73.1 (51.2) | 70.4 (60.7)

8. Primary Outcome: Mean of Number of Doses Administered in Previous Biotherapy
Description: Type of previous biotherapies included were: anti-TNF alpha (infliximab/adalimumab/etanercept/golimumab), selective immuno-suppressant (vedolizumab/abatacept), interleukin inhibitor (anakinra/ustekinumab/tocilizumab), and other. In this outcome measure mean of number of doses administered in previous biotherapy is reported.
Time Frame: Data collected and recorded at study inclusion visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Dose
Arm/Group | Crohn's Disease (CD) | Ulcerative Colitis (UC) | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
Number analyzed (Participants) | 197 | 75 | 55 | 127 | 37
Dose | 38.2 (48.1) | 26.5 (24.5) | 33.5 (30.1) | 39.2 (55.6) | 24.3 (26.6)

9. Primary Outcome: Last Dosage Administered of a Previous Biotherapy
Description: Type of previous biotherapies included were: anti-TNF alpha (infliximab/adalimumab/etanercept/golimumab), selective immuno-suppressant (vedolizumab/abatacept), interleukin inhibitor (anakinra/ustekinumab/tocilizumab), and other. In this outcome measure mean of last dosage (in units) of previous biotherapy administered dose is reported.
Time Frame: Data collected and recorded at study inclusion visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Crohn's Disease (CD) | Ulcerative Colitis (UC) | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
Number analyzed (Participants) | 299 | 124 | 94 | 275 | 59
Units | 104.4 (193.3) | 86.8 (127.2) | 204.8 (255.5) | 216.7 (218.0) | 238.4 (227.9)

10. Primary Outcome: Number of Participants Who Received Concomitant Treatments Prior to Initiation of Inflectra
Description: Following concomitant treatments were received by participants before initiation of Inflectra: 1) Corticosteroids, 2) Salicylates, and 3) Azathioprine/6-MP, Methotrexate, and Cyclosporine.
Time Frame: Data collected and recorded at study inclusion visit
Population: Analysis population included all enrolled participants treated with Inflectra.
Measure: Count of Participants; unit: Participants
Arm/Group | Crohn's Disease (CD) | Ulcerative Colitis (UC) | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
Number analyzed (Participants) | 547 | 230 | 142 | 411 | 96
Participants
  Corticosteroids: Missing | 5 | 1 | 0 | 0 | 0
  Corticosteroids: No | 440 | 162 | 83 | 373 | 82
  Corticosteroids: Yes | 102 | 67 | 59 | 38 | 14
  Salicylates: Missing | 6 | 1 | 0 | 1 | 0
  Salicylates: No | 339 | 70 | 131 | 359 | 90
  Salicylates: Yes | 202 | 159 | 11 | 51 | 6
  Azathioprine/6-MP; Methotrexate; Cyclosporine: Missing | 5 | 1 | 0 | 0 | 0
  Azathioprine/6-MP; Methotrexate; Cyclosporine: No | 144 | 62 | 17 | 224 | 22
  Azathioprine/6-MP; Methotrexate; Cyclosporine: Yes | 398 | 167 | 125 | 187 | 74

11. Secondary Outcome: Physician Global Assessment (PGA) of Disease for RA, SpA and PA
Description: PGA was evaluated in participants with RA, SpA and PA on a 0 to 10 centimeter (cm) visual analog scale (VAS), with 0 cm = no disease activity and 10 cm = worst disease activity possible. Higher scores indicated worse condition.
Time Frame: 24 months
Population: Analysis population included all enrolled participants treated with Inflectra. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure. Analysis for this outcome measure was planned for participants with indications RA, SpA and PA and not for participants with CD and UC.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
Number analyzed (Participants) | 116 | 322 | 76
cm | 3.5 (2.6) | 3.2 (2.4) | 3.2 (2.3)

12. Secondary Outcome: Mean Administered Dose of Inflectra (in mg)
Description: Mean dose (in milligrams [mg]) administered was sum of dose of all infusions administered divided by total number of doses administered.
Time Frame: Inclusion visit up to 6-Month visit, 6-Month visit to 12-Month visit, 12-Month visit up to 18-Month visit, and 18-Month visit up to 24-Month visit
Population: Analysis population included all enrolled participants treated with Inflectra. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable for the specified rows.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Crohn's Disease (CD) | Ulcerative Colitis (UC) | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
Number analyzed (Participants) | 486 | 201 | 119 | 352 | 88
mg
  Inclusion to Month 6 | 451.0 (184.5) | 493.9 (202.1) | 313.7 (125.4) | 406.9 (113.4) | 440.8 (142.5)
  Month 6 to Month 12: number analyzed (Participants) | 437 | 162 | 103 | 314 | 78
  Month 6 to Month 12 | 473.4 (195.6) | 534.0 (213.2) | 313.4 (127.3) | 411.3 (123.0) | 441.2 (152.2)
  Month 12 to Month 18: number analyzed (Participants) | 373 | 133 | 89 | 285 | 73
  Month 12 to Month 18 | 503.1 (211.7) | 520.8 (212.7) | 313.1 (121.7) | 414.8 (120.6) | 437.7 (155.1)
  Month 18 to Month 24: number analyzed (Participants) | 330 | 119 | 78 | 253 | 65
  Month 18 to Month 24 | 515.6 (223.6) | 533.6 (218.5) | 317.5 (109.2) | 417.3 (127.0) | 433.7 (155.6)

13. Secondary Outcome: Mean Administered Posology of Inflectra (in mg/kg)
Description: Mean posology administered was sum of posology of all infusions administered divided by total number of infusions administered. Posology = dose (mg) / weight (kg).
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Crohn's Disease (CD) | Ulcerative Colitis (UC) | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
Number analyzed (Participants) | 486 | 201 | 114 | 334 | 82
mg/kg
  Inclusion to Month 6 | 6.6 (2.2) | 7.0 (2.2) | 4.3 (1.4) | 5.3 (1.1) | 5.4 (1.1)
  Month 6 to Month 12: number analyzed (Participants) | 437 | 162 | 101 | 304 | 75
  Month 6 to Month 12 | 6.8 (2.2) | 7.3 (2.3) | 4.4 (1.4) | 5.4 (1.3) | 5.5 (1.3)
  Month 12 to Month 18: number analyzed (Participants) | 374 | 133 | 88 | 278 | 71
  Month 12 to Month 18 | 7.1 (2.3) | 7.2 (2.4) | 4.4 (1.4) | 5.5 (1.3) | 5.4 (1.3)
  Month 18 to Month 24: number analyzed (Participants) | 331 | 119 | 77 | 249 | 64
  Month 18 to Month 24 | 7.3 (2.3) | 7.4 (2.4) | 4.5 (1.3) | 5.5 (1.3) | 5.4 (1.3)

14. Secondary Outcome: Cumulative Dose
Description: Cumulative dose is the sum of doses administered during inclusion visit to month 6, 12, 18, and 24.
Time Frame: Inclusion visit up to 6-Month visit, Inclusion visit up to 12-Month visit, Inclusion visit up to 18-Month visit, and Inclusion visit up to 24-Month visit
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Crohn's Disease (CD) | Ulcerative Colitis (UC) | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
Number analyzed (Participants) | 486 | 201 | 119 | 352 | 88
mg
  Inclusion to Month 6 | 1028.9 (782.1) | 1071.6 (810.0) | 630.7 (449.0) | 986.1 (589.4) | 1015.4 (832.1)
  Inclusion to Month 12: number analyzed (Participants) | 437 | 162 | 103 | 314 | 78
  Inclusion to Month 12 | 1353.9 (1057.4) | 1437.6 (1118.1) | 804.5 (603.3) | 1202.0 (755.0) | 1251.4 (914.9)
  Inclusion to Month 18: number analyzed (Participants) | 373 | 133 | 89 | 285 | 73
  Inclusion to Month 18 | 1445.2 (1116.0) | 1433.6 (1090.3) | 762.8 (592.4) | 1159.5 (726.7) | 1258.2 (965.2)
  Inclusion to Month 24: number analyzed (Participants) | 330 | 119 | 78 | 253 | 65
  Inclusion to Month 24 | 1718.0 (1305.8) | 1616.9 (1229.6) | 929.6 (668.2) | 1405.8 (892.1) | 1502.0 (1213.7)

15. Secondary Outcome: Mean Infusion Time
Description: Mean infusion time was sum of duration of all infusions administered divided by total number of infusion times administered.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Crohn's Disease (CD) | Ulcerative Colitis (UC) | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
Number analyzed (Participants) | 447 | 183 | 113 | 337 | 85
Minutes
  Inclusion to Month 6 | 75.3 (25.2) | 79.7 (28.0) | 94.8 (30.3) | 92.7 (27.4) | 100.1 (26.4)
  Month 6 to Month 12: number analyzed (Participants) | 403 | 149 | 97 | 301 | 75
  Month 6 to Month 12 | 73.2 (25.1) | 73.9 (29.4) | 88.4 (28.1) | 89.3 (25.9) | 96.8 (29.3)
  Month 12 to Month 18: number analyzed (Participants) | 345 | 121 | 82 | 267 | 68
  Month 12 to Month 18 | 72.7 (25.6) | 70.5 (26.4) | 86.1 (26.3) | 87.6 (25.7) | 94.9 (30.9)
  Month 18 to Month 24: number analyzed (Participants) | 305 | 109 | 69 | 234 | 62
  Month 18 to Month 24 | 71.9 (24.7) | 69.9 (25.0) | 86.9 (26.2) | 87.4 (24.9) | 95.1 (24.1)

16. Secondary Outcome: Mean Time Between Infusions
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Crohn's Disease (CD) | Ulcerative Colitis (UC) | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
Number analyzed (Participants) | 422 | 160 | 101 | 302 | 73
Weeks
  Inclusion to Month 6: number analyzed (Participants) | 340 | 129 | 73 | 251 | 60
  Inclusion to Month 6 | 7.5 (3.5) | 7.7 (3.5) | 7.5 (2.0) | 7.0 (1.7) | 7.2 (1.6)
  Month 6 to Month 12 | 11.9 (8.0) | 13.3 (10.3) | 12.7 (7.3) | 10.7 (6.9) | 11.7 (7.8)
  Month 12 to Month 18: number analyzed (Participants) | 370 | 132 | 88 | 282 | 71
  Month 12 to Month 18 | 12.8 (9.0) | 13.8 (9.8) | 13.7 (8.6) | 12.7 (8.9) | 13.0 (8.7)
  Month 18 to Month 24: number analyzed (Participants) | 255 | 119 | 79 | 253 | 65
  Month 18 to Month 24 | 8.7 (6.2) | 14.4 (11.6) | 15.4 (9.9) | 13.8 (10.4) | 13.3 (8.9)

17. Secondary Outcome: Mean Duration of Post-infusion Monitoring at the Hospital
Description: Mean post-infusion monitoring at hospital was sum of duration of all monitoring at hospital divided by total number monitoring times.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Crohn's Disease (CD) | Ulcerative Colitis (UC) | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
Number analyzed (Participants) | 431 | 177 | 112 | 318 | 80
Minutes
  Inclusion to Month 6 | 53.9 (31.2) | 55.0 (33.5) | 63.6 (30.4) | 66.6 (34.6) | 66.3 (47.1)
  Month 6 to Month 12: number analyzed (Participants) | 386 | 136 | 94 | 287 | 70
  Month 6 to Month 12 | 48.2 (27.9) | 47.3 (26.8) | 55.7 (27.1) | 60.0 (29.1) | 58.7 (37.6)
  Month 12 to Month 18: number analyzed (Participants) | 313 | 105 | 79 | 258 | 64
  Month 12 to Month 18 | 45.9 (23.0) | 45.5 (23.3) | 53.6 (28.8) | 59.1 (30.5) | 54.6 (30.8)
  Month 18 to Month 24: number analyzed (Participants) | 272 | 91 | 69 | 227 | 57
  Month 18 to Month 24 | 48.4 (25.5) | 48.0 (29.6) | 53.8 (31.8) | 58.6 (31.5) | 57.1 (33.3)

18. Secondary Outcome: Absolute Variation in Mean Disease Activity Score (DAS) 28 Compared With Baseline at Month 6, 12, 18, and 24
Description: DAS28 score was evaluated in participants with RA and PA. DAS28 is calculated from the number of swollen joints (SJC) and painful joints (PJC) using the 28 joints count, the erythrocyte sedimentation rate (ESR) (in millimeters per hour [mm/hour]) and participant's global assessment (PtGA) of disease activity (participant rated arthritis activity assessment with scores ranging 0 to 10; higher scores indicated high disease activity). DAS28 was calculated as 0.56 sqrt (DAS 28 tender joint count) + 0.28 sqrt (DAS 28 swollen joint count) + 0.70 ln(ESR [mm/first hour] + 0.014 (PtGA [mm]). Total score range: 0-9.4. DAS 28 score <=2.6 indicated "remission in disease", score between >2.6 and <=3.2 indicated "mildly active disease", score between >3.2 and <=2.6 indicated "moderately active disease", and score >5.1 indicated "very active disease". Absolute variation = mean result of laboratory test during period in question - result of laboratory test at baseline.
Time Frame: Baseline (Inclusion Visit), Month 6, 12, 18, and 24
Population: Analysis population included all enrolled participants treated with Inflectra. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable for the specified rows. Analysis for this outcome measure was planned for participants with indications RA, PA and not for participants with SpA, CD, UC.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rheumatoid Arthritis (RA) | Psoriatic Arthritis (PA)
Number analyzed (Participants) | 95 | 58
Units on a scale
  Month 6 | -0.1 (0.9) | -0.2 (1.1)
  Month 12: number analyzed (Participants) | 83 | 56
  Month 12 | -0.2 (1.1) | -0.3 (1.1)
  Month 18: number analyzed (Participants) | 73 | 54
  Month 18 | -0.2 (1.3) | -0.2 (1.2)
  Month 24: number analyzed (Participants) | 67 | 49
  Month 24 | -0.1 (1.3) | -0.1 (1.4)

19. Secondary Outcome: Absolute Variation in Mean Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Score Compared With Baseline at Month 6, 12, 18, and 24
Description: BASDAI is a set of 6 questions to determine disease activity in participant with SpA. Participants answered each 6 questions on a scale of 0 (no problem) to 10 (the worst problem). The BASDAI score is calculated by computing the mean of questions 5 and 6 and adding it to the sum of questions (Q) 1-4. This score is then divided by 5. BASDAI score = (Q1 + Q2 + Q3+ Q4+ [Q5 + Q6/2])/5. BASDAI score ranges from 0 (best) to 10 (worst), where higher scores meant worse condition. BASDAI score >4 indicated "SpA active", and score <=4 indicated "SpA inactive". Absolute variation = mean result of laboratory test during period in question - result of laboratory test at baseline.
Time Frame: Baseline (Inclusion Visit), Month 6, 12, 18, and 24
Population: Analysis population included all enrolled participants treated with Inflectra. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable for the specified rows. Analysis for this outcome measure was planned for participants with indications SpA and not for participants with RA, PA, CD and UC.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ankylosing Spondylitis (SpA)
Number analyzed (Participants) | 277
Units on a scale
  Month 6 | -0.1 (1.7)
  Month 12: number analyzed (Participants) | 252
  Month 12 | -0.2 (1.7)
  Month 18: number analyzed (Participants) | 235
  Month 18 | -0.2 (1.8)
  Month 24: number analyzed (Participants) | 208
  Month 24 | -0.3 (2.0)

20. Secondary Outcome: Absolute Variation in Mean Bath Ankylosing Spondylitis Functional Index (BASFI) Score Compared With Baseline at Month 6, 12, 18, and 24
Description: BASFI is a set of 10 questions to determine degree of functional limitation in participants with SpA. Participants answered each 10 questions on a scale of 0 (no functional impairment) to 10 (maximal impairment). BASFI score was calculated as mean of scores from 10 questions. BASFI score ranged from 0 (no functional impairment) to 10 (maximal impairment), where higher scores meant worse condition. Score >4 indicated "significant functional impairment", and score <=4 indicated "mild functional impairment". Absolute variation = mean result of laboratory test during period in question - result of laboratory test at baseline.
Time Frame: Baseline (Inclusion Visit), Month 6, 12, 18, and 24
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ankylosing Spondylitis (SpA)
Number analyzed (Participants) | 143
Units on a scale
  Month 6 | -0.1 (1.4)
  Month 12: number analyzed (Participants) | 142
  Month 12 | -0.2 (1.6)
  Month 18: number analyzed (Participants) | 142
  Month 18 | -0.0 (1.8)
  Month 24: number analyzed (Participants) | 117
  Month 24 | 0.1 (1.9)

21. Secondary Outcome: Absolute Variation in Mean Mayo Score Compared With Baseline at Month 6, 12, 18, and 24
Description: Mayo score was evaluated in participants with UC. Mayo score consists of 4 items (stool frequency, rectal bleeding, findings of endoscopy, physician global assessment), each graded from 0 (no severity) to 3 (maximum severity), with higher scores indicating more severe disease. Total score was sum of 4 items resulting in a score range of 0 (no severity) to 12 (maximum severity), where higher score indicated increased severity. Score <=2 indicated "UC inactive", score between >=3 and <=5 indicated "mild UC", score between >=6 and <=10 indicated "moderate UC", and score >11 indicated "severe UC". Absolute variation = mean result of laboratory test during period in question - result of laboratory test at baseline.
Time Frame: Baseline (Inclusion Visit), Month 6, 12, 18, and 24
Population: Analysis population included all enrolled participants treated with Inflectra. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable for the specified rows. Analysis for this outcome measure was planned for participants with indications UC and not for participants with RA, PA, SpA and CD.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ulcerative Colitis (UC)
Number analyzed (Participants) | 66
Units on a scale
  Month 6 | -0.7 (2.3)
  Month 12: number analyzed (Participants) | 46
  Month 12 | -1.3 (2.6)
  Month 18: number analyzed (Participants) | 41
  Month 18 | -1.2 (3.3)
  Month 24: number analyzed (Participants) | 28
  Month 24 | -1.4 (2.9)

22. Secondary Outcome: Absolute Variation in Mean Pediatric Ulcerative Colitis Activity Index (PUCAI) Score Compared With Baseline at Month 6, 12, 18, and 24
Description: PUCAI score was intended for pediatric participants with UC. PUCAI had 6 items with scores as: abdominal pain (no pain =0, pain can be ignored =5, pain cannot be ignored =10); rectal bleeding (none =0, small amount only [in less than 50% of stools] =10, small amount with most stools =20, large amount [>50% of the stool content] =30); stool consistency of most stools (formed =0, partially formed =5, completely unformed =10); number of stools per 24 hours (0-2 =0, 3-5 =5, 6-8 =10, >8 =15); nocturnal stools (no =0, yes =10); activity level (no limitation of activity =0, occasional limitation of activity =5, severely restricted activity =10). PUCAI score = sum of scores of 6 items; score range of 0= no severity to 85= extreme severity. PUCAI score <10: UC in remission, score between >=10 and <35: mild UC, score between >=35 and <65: moderate UC, and score >=65: severe UC. Absolute variation = mean result of laboratory test during period in question - result of laboratory test at baseline.
Time Frame: Baseline (Inclusion Visit), Month 6, 12, 18, and 24
Population: Analysis population included all enrolled participants treated with Inflectra. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable for the specified rows. Analysis for this outcome measure was planned for pediatric participants with indications UC and not for participants with RA, PA, SpA and CD.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ulcerative Colitis (UC)
Number analyzed (Participants) | 7
Units on a scale
  Month 6 | -5.3 (22.6)
  Month 12: number analyzed (Participants) | 6
  Month 12 | 2.2 (6.8)
  Month 18: number analyzed (Participants) | 5
  Month 18 | 1.8 (5.4)
  Month 24: number analyzed (Participants) | 4
  Month 24 | 2.2 (6.0)

23. Secondary Outcome: Absolute Variation in Mean Colitis Endoscopic Index of Severity (UCEIS) Score Compared With Baseline at Month 6, 12, 18, and 24
Description: UCEIS score was evaluated in participants with indication UC. It had 3 sub-scales: endoscopic vascular pattern (scored 0 [normal pattern] to 2 [complete obliteration of vascular pattern]), bleeding (scored 0 [none] to 3 [luminal moderate or severe]), erosions and ulcerations (scored 0 [none] to 3 [deep ulcers]). UCEIS total score was calculated by sum of all 3 sub-scale scores. Total score ranged from 0 (remission in disease) to 8 (extreme severity of disease), with higher scores indicating more severe disease. Absolute variation = mean result of laboratory test during period in question - result of laboratory test at baseline.
Time Frame: Baseline (Inclusion Visit), Month 6, 12, 18, and 24
Population: Analysis population included all enrolled participants treated with Inflectra. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable for the specified rows. Analysis for this outcome measure was planned for participants with indications UC and not for participants with RA, SpA, PA and CD.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ulcerative Colitis (UC)
Number analyzed (Participants) | 12
Units on a scale
  Month 6 | 0.25 (4.20)
  Month 12: number analyzed (Participants) | 10
  Month 12 | -0.80 (3.71)
  Month 18: number analyzed (Participants) | 8
  Month 18 | 0.00 (2.62)
  Month 24: number analyzed (Participants) | 4
  Month 24 | -2.50 (2.38)

24. Secondary Outcome: Absolute Variation in Mean Harvey-Bradshaw Score Compared With Baseline at Month 6, 12, 18, and 24
Description: Harvey-Bradshaw score was evaluated for indication CD. Harvey-Bradshaw measures 5 parameters; general well-being (0= very well to 4= terrible), abdominal pain (0= none to 3= severe), number of liquid stools per day (0 to no maximum score), presence of an abdominal mass on physical exam (0= none to 3= definite and tender), and whether there are any complications (0= no complications, 1= arthralgia, 2= uveitis, 3= erythema nodosum, 4= aphthous ulcer, 5= pyoderma gangrenosum, 6= anal fissure, 7= new fistula, 8= abscess). Total HBI score: sum of all 5 individual parameters, minimum score is 0 and there was no pre-specified maximum score as it depended on number of liquids stools. Higher HBI scores = greater disease activity score <4 indicated "Inactive disease", score >=4 and/or <=12 indicated "Active disease", and score >12 indicated "Very active disease". Absolute variation = mean result of laboratory test during period in question - result of laboratory test at baseline.
Time Frame: Baseline (Inclusion Visit), Month 6, 12, 18, and 24
Population: Analysis population included all enrolled participants treated with Inflectra. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable for the specified rows. Analysis for this outcome measure was planned for participants with indications CD and not for participants with RA, SpA, PA, UC.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Crohn's Disease (CD)
Number analyzed (Participants) | 322
Units on a scale
  Month 6 | -0.1 (2.4)
  Month 12: number analyzed (Participants) | 286
  Month 12 | -0.2 (2.3)
  Month 18: number analyzed (Participants) | 239
  Month 18 | -0.4 (2.2)
  Month 24: number analyzed (Participants) | 210
  Month 24 | -0.6 (2.5)

25. Secondary Outcome: Absolute Variation in Mean Crohn's Disease Endoscopic Index of Severity (CDEIS) Score Compared With Baseline at Month 6, 12, 18, and 24
Description: CDEIS is an index for determining the severity of CD with endoscopic localization to ileum and colon. CDEIS considered 4 parameters: deep ulcerations, superficial ulcerations, ulcerated and non-ulcerated surface, and the presence of ulcerated/non-ulcerated stenosis. These 4 parameters were evaluated in 5 pre-defined segments of the colon (ileum, ascending colon, transverse colon, descending colon and sigmoid loop, and rectum). CDEIS score ranged from 0 (no lesions) to 44 (severe lesions) where higher scores indicate more severity. CDEIS score <=7 indicated "Endoscopic remission", and score >7 indicated "Absence of endoscopic remission". Absolute variation = mean result of laboratory test during period in question - result of laboratory test at baseline.
Time Frame: Baseline (Inclusion Visit), Month 6, 12, 18, and 24
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Crohn's Disease (CD)
Number analyzed (Participants) | 12
Units on a scale
  Month 6: number analyzed (Participants) | 7
  Month 6 | -2.35 (4.03)
  Month 12 | -5.98 (7.40)
  Month 18: number analyzed (Participants) | 3
  Month 18 | -1.37 (1.50)
  Month 24: number analyzed (Participants) | 0

26. Secondary Outcome: Absolute Variation of Mean Global Disease Assessment Compared With Baseline at Month 6, 12, 18, and 24
Description: The global disease assessment by the physician for participants with RA, SpA and PA was evaluated on a 0 to 10 cm VAS, with 0 cm = no disease activity and 10 cm = worst disease activity. Higher scores indicated worse condition. Absolute variation = mean result of laboratory test during period in question - result of laboratory test at baseline.
Time Frame: Baseline (Inclusion Visit), Month 6, 12, 18, and 24
Population: Analysis population included all enrolled participants treated with Inflectra. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable for the specified rows. Analysis for this outcome measure was planned for participants with indications RA, SpA, PA and not for participants with CD, UC.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
Number analyzed (Participants) | 75 | 192 | 54
Units on a scale
  Month 6: number analyzed (Participants) | 75 | 179 | 45
  Month 6 | -0.3 (2.3) | -0.0 (2.2) | -0.5 (2.2)
  Month 12: number analyzed (Participants) | 69 | 192 | 54
  Month 12 | -0.4 (2.5) | -0.2 (2.3) | -0.4 (2.3)
  Month 18: number analyzed (Participants) | 61 | 174 | 45
  Month 18 | -0.5 (2.5) | -0.1 (2.2) | -0.3 (2.4)
  Month 24: number analyzed (Participants) | 53 | 173 | 39
  Month 24 | 0.1 (3.1) | -0.1 (2.4) | -0.5 (2.6)

27. Secondary Outcome: Absolute Variation of Mean Fatigue Score Compared With Baseline at Month 6, 12, 18, and 24
Description: Fatigue score was evaluated among participants with RA, SpA, and PA. Participants' fatigue severity was measured on a VAS with a score range of 0 (no fatigue) to 10 (highest level of fatigue). Higher score signifies more severity. Absolute variation = mean result of laboratory test during period in question - result of laboratory test at baseline.
Time Frame: Baseline (Inclusion Visit), Month 6, 12, 18, and 24
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
Number analyzed (Participants) | 69 | 241 | 50
Units on a scale
  Month 6: number analyzed (Participants) | 69 | 223 | 43
  Month 6 | -0.6 (1.8) | 0.0 (2.2) | -0.4 (2.1)
  Month 12: number analyzed (Participants) | 67 | 241 | 50
  Month 12 | 0.1 (2.7) | 0.1 (2.3) | -0.3 (2.2)
  Month 18: number analyzed (Participants) | 57 | 215 | 45
  Month 18 | -0.3 (2.2) | -0.1 (2.3) | 0.1 (2.6)
  Month 24: number analyzed (Participants) | 50 | 184 | 40
  Month 24 | 0.0 (2.2) | -0.1 (2.6) | 0.4 (2.5)

28. Secondary Outcome: Absolute Variation in Mean Simple Disease Activity Index (SDAI) Score Compared With Baseline at Month 6, 12, 18, and 24
Description: SDAI was evaluated in participants with indication RA. SDAI is the numerical sum of 5 parameters: TJC and SJC based on a 28-joint assessment, PtGA and PGA assessed on 0 (very well) -10 cm (worst) VAS; higher scores = greater affection due to disease activity, and C-reactive protein (CRP) (mg/dL). SDAI total score =0 (no disease) to 86 (extreme severity of disease), where higher scores indicated higher disease activity. SDAI score <=3.3 indicated "achievement of remission state", score >3.3 and/or <=11 indicated "mildly active state", score >11 and/or <=26 indicated "moderately active state", and score >26 indicated "very active state". Absolute variation = mean result of laboratory test during period in question - result of laboratory test at baseline.
Time Frame: Baseline (Inclusion Visit), Month 6, 12, 18, and 24
Population: Analysis population included all enrolled participants treated with Inflectra. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable for the specified rows. Analysis for this outcome measure was planned for participants with indication RA, and not for participants with SpA, PA, CD, UC.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rheumatoid Arthritis (RA)
Number analyzed (Participants) | 54
Units on a scale
  Month 6 | -1.6 (10.7)
  Month 12: number analyzed (Participants) | 52
  Month 12 | -1.5 (11.4)
  Month 18: number analyzed (Participants) | 53
  Month 18 | -4.0 (14.0)
  Month 24: number analyzed (Participants) | 45
  Month 24 | -3.1 (11.9)

29. Secondary Outcome: Absolute Variation in Mean Health Assessment Questionnaire (HAQ) Score Compared With Baseline at Month 6, 12, 18, and 24
Description: HAQ score was evaluated for indication RA. HAQ assesses degree of difficulty participant had experienced during past week in 8 domains of daily activities: dressing & grooming, arising, eating, walking, hygiene, reach, grip and other activities. For each question in questionnaire, level of difficulty was scored from 0 (no difficulty) to 3 (unable to do). Any activity requiring assistance from another individual or required use of assistive device would adjust to minimum score of 2 to represent more limited functional status. Overall score = sum of scores divided by number of domains answered. Total possible score range was 0 (no difficulty) to 3 (unable to do). Higher score = more difficulty in performing daily living activities. HAQ score >0.5 indicated "Existence of functional disability" & HAQ score <=0.5 indicated "Absence of functional disability". Absolute variation = mean result of laboratory test during period in question - result of laboratory test at baseline.
Time Frame: Baseline (Inclusion Visit), Month 6, 12, 18, and 24
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rheumatoid Arthritis (RA)
Number analyzed (Participants) | 15
Units on a scale
  Month 6: number analyzed (Participants) | 5
  Month 6 | -0.3 (0.1)
  Month 12 | 0.0 (0.4)
  Month 18: number analyzed (Participants) | 10
  Month 18 | -0.2 (0.5)
  Month 24: number analyzed (Participants) | 4
  Month 24 | 0.4 (0.6)

30. Secondary Outcome: Absolute Variation in Mean Ankylosing Spondylitis Disease Activity Score (ASDAS) Score Compared With Baseline at Month 6, 12, 18, and 24
Description: ASDAS score was evaluated for indication SpA. It is a score combining the assessment of overall pain (Q1), duration of morning stiffness (Q2), peripheral pain/swelling (Q3), PtGA (assessed on a sale of 0 [not active] to 10 [very active]), and CRP in mg/L. ASDAS total score ranged from 0 (no disease) to 10 (maximum severity), higher score indicates greater severity of disease and was derived using the following formula: ASDAS =0.12*Q1 + 0.06*Q2 + 0.11* PtGA + 0.07*Q3 + 0.58*ln (CRP+1). ASDAS score <1.3 indicated "SpA inactive", ASDAS score >=1.3 and/or <2.1 indicated "SpA mildly active", ASDAS score >=2.1 and/or <=3.5 indicated "SpA moderately active", and ASDAS score >3.5 indicated "SpA very active". Absolute variation = mean result of laboratory test during period in question - result of laboratory test at baseline.
Time Frame: Baseline (Inclusion Visit), Month 6, 12, 18, and 24
Population: Analysis population included all enrolled participants treated with Inflectra. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable for the specified rows. Analysis for this outcome measure was planned for participants with indication SpA, and not for participants with RA, PA, CD, UC.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ankylosing Spondylitis (SpA)
Number analyzed (Participants) | 135
Units on a scale
  Month 6: number analyzed (Participants) | 131
  Month 6 | -0.1 (0.7)
  Month 12 | -0.1 (0.7)
  Month 18: number analyzed (Participants) | 130
  Month 18 | -0.2 (0.9)
  Month 24: number analyzed (Participants) | 106
  Month 24 | -0.2 (0.8)

31. Secondary Outcome: Cook and Medley Score at Baseline
Description: Cook-Medley questionnaire, also called cynical distrust scale, contained 8 items, scoring from 0 (trust) to 4 (no trust). The total score of the questionnaire was calculated by adding together the scores for the 8 items. Total possible score range was from 0 (trust) to 32 (no trust), higher score signifies greater cynical distrust. This outcome measure was evaluated in participants who were informed of a switch from infliximab reference to Inflectra.
Time Frame: Baseline (data recorded at inclusion visit)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Crohn's Disease (CD) | Ulcerative Colitis (UC) | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
Number analyzed (Participants) | 186 | 61 | 66 | 185 | 41
Units on a scale | 19.0 (4.9) | 17.1 (5.7) | 18.7 (4.1) | 18.1 (5.1) | 20.0 (6.1)

32. Secondary Outcome: Stress Score
Description: The questionnaire on stress after the switch to the biosimilar contained 3 items (emotional reactivity, repetition syndrome and tendency to avoid), each scored from 0 (no stress) to 4 (extreme stress). The overall score of stress was calculated by adding together the scores for the 3 items, ranged from 0 (no stress) to 12 (highest level of stress), higher scores indicated greater levels of stress. This outcome measure was evaluated in participants who were informed of a switch from infliximab reference to Inflectra.
Time Frame: Baseline (inclusion visit) up to Month 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Crohn's Disease (CD) | Ulcerative Colitis (UC) | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
Number analyzed (Participants) | 186 | 61 | 66 | 185 | 41
Units on a scale | 2.3 (1.7) | 2.0 (2.6) | 1.3 (1.6) | 1.9 (2.1) | 3.4 (2.7)

33. Secondary Outcome: General Anxiety Disorder (GAD7) Score
Description: GAD7: questionnaire of anxiety with 7 items, scoring from 0 (no anxiety) to 3 (extreme anxiety). The total GAD7 score was calculated by adding together the scores for the 7 items, ranged from 0 (no anxiety) to 21 (extreme anxiety), higher scores indicated severe anxiety. This outcome measure was evaluated in participants who were informed of a switch from infliximab reference to Inflectra.
Time Frame: Baseline (inclusion visit) through post each infusion (during 2 years)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Crohn's Disease (CD) | Ulcerative Colitis (UC) | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
Number analyzed (Participants) | 186 | 61 | 66 | 185 | 41
Units on a scale | 5.5 (3.7) | 3.4 (3.2) | 3.8 (5.1) | 4.8 (5.1) | 7.8 (6.3)

34. Secondary Outcome: Number of Participants With Immunogenicity Assay at Inclusion Visit
Time Frame: Baseline (data recorded at inclusion visit)
Population: Analysis population included all enrolled participants treated with Inflectra.
Measure: Count of Participants; unit: Participants
Arm/Group | Crohn's Disease (CD) | Ulcerative Colitis (UC) | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
Number analyzed (Participants) | 547 | 230 | 142 | 411 | 96
Participants | 87 | 44 | 13 | 24 | 5

35. Secondary Outcome: Number of Participants With Anti-Infliximab Antibody Assay Assessment at Inclusion Visit
Time Frame: Baseline (data recorded at inclusion visit)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Crohn's Disease (CD) | Ulcerative Colitis (UC) | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
Number analyzed (Participants) | 87 | 44 | 13 | 24 | 5
Participants | 79 | 37 | 9 | 24 | 5

36. Secondary Outcome: Number of Participants With Presence of Anti-infliximab Antibodies at Inclusion Visit
Time Frame: Baseline (data recorded at inclusion visit)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Crohn's Disease (CD) | Ulcerative Colitis (UC) | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
Number analyzed (Participants) | 79 | 37 | 9 | 24 | 5
Participants | 9 | 6 | 1 | 8 | 3

37. Secondary Outcome: Number of Participants With Infliximab Trough Level (IFX-TL) Assay at Inclusion Visit
Description: Trough level was plasma concentration of drug before infusion.
Time Frame: Baseline (data recorded at inclusion visit)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Crohn's Disease (CD) | Ulcerative Colitis (UC) | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
Number analyzed (Participants) | 87 | 44 | 13 | 24 | 5
Participants | 82 | 40 | 8 | 21 | 5

38. Secondary Outcome: Infliximab Trough Level (IFX-TL) at Inclusion Visit
Description: Trough level was plasma concentration of drug before infusion.
Time Frame: Before infusion at baseline (data recorded at inclusion visit)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Crohn's Disease (CD) | Ulcerative Colitis (UC) | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
Number analyzed (Participants) | 82 | 40 | 8 | 21 | 5
micrograms per milliliter | 6.69 (5.58) | 7.66 (5.94) | 6.06 (6.83) | 7.32 (6.14) | 7.40 (2.82)

39. Secondary Outcome: Mean of Number of Immunogenicity Assays Done (Inclusion Visit up to 6-Month Visit, 6-Month Visit up to 12-Month Visit, 12-Month Visit up to 18-Month Visit, and 18-Month Visit up to 24-Month Visit)
Time Frame: Inclusion visit up to 6-Month visit, 6-Month visit up to 12-Month visit, 12-Month visit up to 18-Month visit, and 18-Month visit up to 24-Month visit
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Assays
Arm/Group | Crohn's Disease (CD) | Ulcerative Colitis (UC) | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
Number analyzed (Participants) | 486 | 198 | 118 | 354 | 88
Assays
  Inclusion up to Month 6 | 0.3 (0.8) | 0.4 (0.8) | 0.1 (0.3) | 0.1 (0.3) | 0.1 (0.3)
  Month 6 to Month 12: number analyzed (Participants) | 434 | 162 | 102 | 315 | 78
  Month 6 to Month 12 | 0.5 (1.0) | 0.4 (1.0) | 0.1 (0.3) | 0.1 (0.4) | 0.1 (0.3)
  Month 12 to Month 18: number analyzed (Participants) | 372 | 134 | 88 | 287 | 73
  Month 12 to Month 18 | 0.5 (1.0) | 0.6 (1.1) | 0.1 (0.4) | 0.1 (0.4) | 0.2 (0.4)
  Month 18 to Month 24: number analyzed (Participants) | 331 | 118 | 78 | 253 | 65
  Month 18 to Month 24 | 0.5 (1.2) | 0.6 (1.2) | 0.2 (0.4) | 0.1 (0.3) | 0.1 (0.4)

40. Secondary Outcome: Number of Participants With Presence of At-least 1 Anti-Infliximab Antibodies (Inclusion Visit up to 6-Month Visit, 6-Month Visit up to 12-Month Visit, 12-Month Visit up to 18-Month Visit, and 18-Month Visit up to 24-Month Visit)
Time Frame: as for outcome 39
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Crohn's Disease (CD) | Ulcerative Colitis (UC) | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
Number analyzed (Participants) | 115 | 48 | 14 | 40 | 11
Participants
  Inclusion to Month 6: number analyzed (Participants) | 101 | 48 | 11 | 38 | 9
  Inclusion to Month 6 | 7 | 3 | 4 | 7 | 2
  Month 6 to Month 12: number analyzed (Participants) | 115 | 34 | 12 | 40 | 10
  Month 6 to Month 12 | 5 | 2 | 7 | 9 | 5
  Month 12 to Month 18: number analyzed (Participants) | 95 | 36 | 12 | 27 | 11
  Month 12 to Month 18 | 5 | 5 | 7 | 9 | 5
  Month 18 to Month 24: number analyzed (Participants) | 95 | 30 | 14 | 29 | 7
  Month 18 to Month 24 | 9 | 2 | 7 | 8 | 4

41. Secondary Outcome: Mean Inflectra Trough Level (IFX-TL) (Inclusion Visit up to 6-Month Visit, 6-Month Visit up to 12-Month Visit, 12-Month Visit up to 18-Month Visit, and 18-Month Visit up to 24-Month Visit)
Description: Trough level was plasma concentration of drug before infusion. In this outcome measure mean of all IFX-TLs for all infusions occurring during specified duration is reported.
Time Frame: Before every infusion occurred during: inclusion visit up to 6-Month visit; 6-Month visit up to 12-Month visit; 12-Month visit up to 18-Month visit, and 18-Month visit up to 24-Month visit
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Crohn's Disease (CD) | Ulcerative Colitis (UC) | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
Number analyzed (Participants) | 114 | 45 | 14 | 38 | 11
micrograms per milliliter
  Inclusion to Month 6: number analyzed (Participants) | 100 | 45 | 11 | 36 | 8
  Inclusion to Month 6 | 8.4 (13.1) | 6.5 (5.4) | 4.2 (3.9) | 6.9 (5.9) | 9.2 (6.2)
  Month 6 to Month 12: number analyzed (Participants) | 114 | 34 | 12 | 38 | 10
  Month 6 to Month 12 | 7.3 (7.9) | 7.0 (5.1) | 3.5 (5.3) | 8.9 (6.1) | 7.4 (6.7)
  Month 12 to Month 18: number analyzed (Participants) | 94 | 35 | 11 | 26 | 11
  Month 12 to Month 18 | 7.7 (5.9) | 5.3 (4.2) | 2.3 (3.3) | 7.2 (5.2) | 6.8 (6.0)
  Month 18 to Month 24: number analyzed (Participants) | 94 | 30 | 14 | 28 | 7
  Month 18 to Month 24 | 7.7 (5.5) | 6.8 (4.5) | 2.1 (2.5) | 7.8 (6.4) | 8.5 (6.5)

ADVERSE EVENTS:
Time Frame: During 2 years post inclusion in the study (24 months)
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Crohn's Disease (CD) | Ulcerative Colitis (UC) | Rheumatoid Arthritis (RA) | Ankylosing Spondylitis (SpA) | Psoriatic Arthritis (PA)
All-Cause Mortality (participants affected / at risk) | 1/547 | 2/230 | 1/142 | 0/411 | 0/96
Serious Adverse Events (participants affected / at risk) | 73/547 | 28/230 | 20/142 | 47/411 | 10/96
Other Adverse Events (participants affected / at risk) | 252/547 | 91/230 | 62/142 | 219/411 | 49/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crohn's Disease (CD) (N=547) | Ulcerative Colitis (UC) (N=230) | Rheumatoid Arthritis (RA) (N=142) | Ankylosing Spondylitis (SpA) (N=411) | Psoriatic Arthritis (PA) (N=96)
CROHN'S DISEASE (Gastrointestinal disorders) | 6 | 0 | 0 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 | 1 | 0 | 0 | 0
COLITIS (Gastrointestinal disorders) | 0 | 3 | 0 | 1 | 0
COLITIS ULCERATIVE (Gastrointestinal disorders) | 0 | 4 | 0 | 0 | 0
ILEAL STENOSIS (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0
LARGE INTESTINAL STENOSIS (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
ABDOMINAL RIGIDITY (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
ANAL STENOSIS (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
DISTAL INTESTINAL OBSTRUCTION SYNDROME (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
ENTERITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
ENTEROCOLITIS (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
ENTEROCUTANEOUS FISTULA (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
HIATUS HERNIA (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
INTRA-ABDOMINAL FLUID COLLECTION (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
OESOPHAGITIS ULCERATIVE (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
SALIVARY GLAND PAIN (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
ANAL ABSCESS (Infections and infestations) | 4 | 0 | 0 | 0 | 0
PERITONITIS (Infections and infestations) | 3 | 0 | 0 | 1 | 0
HERPES ZOSTER (Infections and infestations) | 1 | 0 | 2 | 0 | 0
HEPATITIS E (Infections and infestations) | 1 | 0 | 0 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 1
ABDOMINAL ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
ABSCESS INTESTINAL (Infections and infestations) | 1 | 0 | 0 | 0 | 0
ANAL FISTULA INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0
CAMPYLOBACTER INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 0
CYTOMEGALOVIRUS HEPATITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0
ERYSIPELAS (Infections and infestations) | 0 | 0 | 1 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
GASTROINTESTINAL INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0
LEGIONELLA INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0
PELVIC ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
PERINEAL ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
PERIUMBILICAL ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 1 | 0
PNEUMONIA HAEMOPHILUS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
PNEUMONIA LEGIONELLA (Infections and infestations) | 0 | 0 | 0 | 1 | 0
PULMONARY TUBERCULOSIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
PYELONEPHRITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION BACTERIAL (Infections and infestations) | 0 | 0 | 0 | 1 | 0
VISCERAL LEISHMANIASIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0
ILEOCOLOSTOMY (Surgical and medical procedures) | 7 | 0 | 0 | 0 | 0
CANCER SURGERY (Surgical and medical procedures) | 1 | 1 | 0 | 0 | 0
EVENTRATION REPAIR (Surgical and medical procedures) | 2 | 0 | 0 | 0 | 0
GASTRECTOMY (Surgical and medical procedures) | 0 | 0 | 1 | 1 | 0
ABDOMINAL OPERATION (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
ARTHRODESIS (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
CARDIAC RESYNCHRONISATION THERAPY (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
CHOLECYSTECTOMY (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
COLECTOMY TOTAL (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
DRUG DELIVERY DEVICE IMPLANTATION (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
FISTULA REPAIR (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
HIP ARTHROPLASTY (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
HYDROCELE OPERATION (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
ILEOSTOMY (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
KNEE ARTHROPLASTY (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
ORCHIDOPEXY (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
OSTEOSYNTHESIS (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
OSTEOTOMY (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
PROCTECTOMY (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
RIB EXCISION (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
SHOULDER ARTHROPLASTY (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
SIGMOIDECTOMY (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
STOMA CLOSURE (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 2 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0 | 0
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
COLORECTAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
HODGKIN'S DISEASE NODULAR SCLEROSIS STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
INTESTINAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
MALIGNANT MELANOMA IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
PYOGENIC GRANULOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
RECTAL ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
DRUG INEFFECTIVE (General disorders) | 1 | 2 | 1 | 0 | 0
CONDITION AGGRAVATED (General disorders) | 0 | 1 | 0 | 0 | 0
DEATH (General disorders) | 1 | 0 | 0 | 0 | 0 — Family reported about the death of a participant and there was no autopsy or any other information was available. Hence, reason for serious AE term "Death" was unknown.
DISEASE PROGRESSION (General disorders) | 1 | 0 | 0 | 0 | 0
DISEASE RECURRENCE (General disorders) | 0 | 0 | 1 | 0 | 0
HYPERTHERMIA (General disorders) | 1 | 0 | 0 | 0 | 0
INFLAMMATION (General disorders) | 0 | 0 | 0 | 1 | 0
PROLAPSE (General disorders) | 1 | 0 | 0 | 0 | 0
STENOSIS (General disorders) | 1 | 0 | 0 | 0 | 0
THERAPEUTIC RESPONSE SHORTENED (General disorders) | 0 | 0 | 0 | 1 | 0
VASCULAR STENT RESTENOSIS (General disorders) | 0 | 0 | 0 | 0 | 1
FALL (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 0 | 0
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0
ACCIDENT AT WORK (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
ANASTOMOTIC LEAK (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
DRUG ADMINISTRATION ERROR (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
HEAD INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
INJECTION RELATED REACTION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
LUPUS-LIKE SYNDROME (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
ANKYLOSING SPONDYLITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
FISTULA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
INTERVERTEBRAL DISC DISORDER (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
PSORIATIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
SCIATICA (Nervous system disorders) | 0 | 0 | 0 | 2 | 1
AGEUSIA (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
DIZZINESS (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
EPILEPSY (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
FACIAL PARALYSIS (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
HEADACHE (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
MIGRAINE (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
PARKINSON'S DISEASE (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
RADICULOPATHY (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
THALAMUS HAEMORRHAGE (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
CARDIAC FAILURE (Cardiac disorders) | 0 | 2 | 1 | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
CARDIAC FLUTTER (Cardiac disorders) | 0 | 0 | 0 | 2 | 0
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
PERICARDITIS (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
LARYNGEAL CYST (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0
CHOLANGITIS (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
HEPATOCELLULAR INJURY (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
LIVER INJURY (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
PORTAL HYPERTENSION (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
PROSTATITIS (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
DYSMENORRHOEA (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
FEMALE GENITAL TRACT FISTULA (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
TESTICULAR TORSION (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 1 | 2 | 0 | 1 | 0
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
IMMUNE THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
MICROCYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
HYPERSENSITIVITY (Immune system disorders) | 1 | 0 | 1 | 0 | 0
ANAPHYLACTIC SHOCK (Immune system disorders) | 0 | 0 | 1 | 0 | 0
SARCOIDOSIS (Immune system disorders) | 0 | 1 | 0 | 0 | 0
RENAL COLIC (Renal and urinary disorders) | 1 | 0 | 0 | 2 | 0
URINARY RETENTION (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
DACRYOSTENOSIS ACQUIRED (Eye disorders) | 0 | 0 | 0 | 0 | 1
LACRIMATION INCREASED (Eye disorders) | 0 | 0 | 0 | 0 | 1
OCULAR MYASTHENIA (Eye disorders) | 0 | 0 | 0 | 1 | 0
SCLERITIS (Eye disorders) | 0 | 0 | 0 | 1 | 0
PRURIGO (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
PSORIASIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
OBESITY (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
DEPRESSION (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 | 0 | 0 | 1 | 0
PHLEBITIS (Vascular disorders) | 1 | 0 | 0 | 0 | 0
LAPAROSCOPY (Investigations) | 1 | 0 | 0 | 0 | 0
PREGNANCY OF PARTNER (Social circumstances) | 0 | 0 | 0 | 0 | 1
COLECTOMY (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crohn's Disease (CD) (N=547) | Ulcerative Colitis (UC) (N=230) | Rheumatoid Arthritis (RA) (N=142) | Ankylosing Spondylitis (SpA) (N=411) | Psoriatic Arthritis (PA) (N=96)
BRONCHITIS (Infections and infestations) | 16 | 0 | 10 | 25 | 8
NASOPHARYNGITIS (Infections and infestations) | 20 | 2 | 1 | 16 | 4
TONSILLITIS (Infections and infestations) | 19 | 3 | 0 | 14 | 3
RHINITIS (Infections and infestations) | 11 | 1 | 2 | 14 | 1
SINUSITIS (Infections and infestations) | 7 | 3 | 1 | 12 | 5
URINARY TRACT INFECTION (Infections and infestations) | 16 | 1 | 2 | 6 | 3
GASTROENTERITIS (Infections and infestations) | 8 | 2 | 3 | 10 | 0
CONJUNCTIVITIS (Infections and infestations) | 14 | 0 | 0 | 4 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 6 | 1 | 1 | 5 | 1
TOOTH ABSCESS (Infections and infestations) | 5 | 0 | 1 | 3 | 3
EAR INFECTION (Infections and infestations) | 3 | 1 | 0 | 4 | 2
LUNG INFECTION (Infections and infestations) | 2 | 1 | 2 | 3 | 2
HERPES ZOSTER (Infections and infestations) | 4 | 0 | 3 | 1 | 1
INFECTION (Infections and infestations) | 5 | 1 | 0 | 3 | 0
INFLUENZA (Infections and infestations) | 3 | 1 | 2 | 2 | 1
TOOTH INFECTION (Infections and infestations) | 3 | 1 | 0 | 5 | 0
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 | 0 | 0 | 3 | 1
ORAL HERPES (Infections and infestations) | 3 | 1 | 0 | 4 | 0
TRACHEITIS (Infections and infestations) | 2 | 2 | 0 | 4 | 0
CYSTITIS (Infections and infestations) | 2 | 0 | 1 | 1 | 3
FOLLICULITIS (Infections and infestations) | 4 | 1 | 0 | 1 | 1
PHARYNGITIS (Infections and infestations) | 4 | 1 | 0 | 1 | 1
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 1 | 1 | 0 | 4 | 1
VIRAL INFECTION (Infections and infestations) | 2 | 1 | 1 | 2 | 0
ANGULAR CHEILITIS (Infections and infestations) | 5 | 0 | 0 | 0 | 0
ERYSIPELAS (Infections and infestations) | 3 | 0 | 0 | 2 | 0
FUNGAL INFECTION (Infections and infestations) | 2 | 0 | 0 | 2 | 0
GASTROENTERITIS VIRAL (Infections and infestations) | 3 | 1 | 0 | 0 | 0
HERPES SIMPLEX (Infections and infestations) | 2 | 1 | 1 | 0 | 0
DIVERTICULITIS (Infections and infestations) | 0 | 0 | 0 | 2 | 1
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1 | 1 | 0 | 0 | 1
FURUNCLE (Infections and infestations) | 2 | 0 | 0 | 1 | 0
LARYNGITIS (Infections and infestations) | 1 | 0 | 0 | 2 | 0
ONYCHOMYCOSIS (Infections and infestations) | 1 | 0 | 0 | 2 | 0
OTITIS EXTERNA (Infections and infestations) | 0 | 0 | 0 | 3 | 0
SUBCUTANEOUS ABSCESS (Infections and infestations) | 2 | 0 | 0 | 0 | 1
TRACHEOBRONCHITIS (Infections and infestations) | 0 | 0 | 1 | 2 | 0
ANAL FUNGAL INFECTION (Infections and infestations) | 1 | 1 | 0 | 0 | 0
CYSTITIS ESCHERICHIA (Infections and infestations) | 0 | 1 | 0 | 0 | 1
DERMATOPHYTOSIS OF NAIL (Infections and infestations) | 1 | 0 | 0 | 1 | 0
EPSTEIN-BARR VIRUS INFECTION (Infections and infestations) | 1 | 0 | 1 | 0 | 0
GROIN ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0 | 1
HELICOBACTER INFECTION (Infections and infestations) | 1 | 1 | 0 | 0 | 0
HORDEOLUM (Infections and infestations) | 0 | 1 | 0 | 1 | 0
LOCALISED INFECTION (Infections and infestations) | 0 | 1 | 0 | 1 | 0
MASTITIS (Infections and infestations) | 0 | 1 | 0 | 1 | 0
ORAL FUNGAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 1
PERIODONTITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 1
PERITONSILLAR ABSCESS (Infections and infestations) | 2 | 0 | 0 | 0 | 0
PYELONEPHRITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 1
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 | 1 | 0 | 1 | 0
RASH PUSTULAR (Infections and infestations) | 1 | 0 | 1 | 0 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1 | 1 | 0
SKIN INFECTION (Infections and infestations) | 1 | 0 | 0 | 1 | 0
VAGINAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 1
VIRAL PHARYNGITIS (Infections and infestations) | 1 | 0 | 1 | 0 | 0
ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
ABSCESS INTESTINAL (Infections and infestations) | 1 | 0 | 0 | 0 | 0
ABSCESS JAW (Infections and infestations) | 0 | 0 | 0 | 1 | 0
ACARODERMATITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1
ACUTE SINUSITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
ANAL ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
CAMPYLOBACTER INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0
CANDIDA INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0
CHLAMYDIAL INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 0
CONJUNCTIVITIS VIRAL (Infections and infestations) | 0 | 1 | 0 | 0 | 0
CORNEAL ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
CORONA VIRUS INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0
DERMO-HYPODERMITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
ENDOMETRITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
ENTEROCOCCAL INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0
EPIDIDYMITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
FUNGAL SKIN INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0
GARDNERELLA INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0
GASTROINTESTINAL VIRAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0
GENITAL HERPES SIMPLEX (Infections and infestations) | 0 | 0 | 0 | 1 | 0
GENITAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0
GINGIVITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
HELICOBACTER GASTRITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1
HERPES VIRUS INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1
INFECTED DERMAL CYST (Infections and infestations) | 0 | 0 | 0 | 1 | 0
INFECTIOUS MONONUCLEOSIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0
LYMPHANGITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
NASAL HERPES (Infections and infestations) | 1 | 0 | 0 | 0 | 0
OPHTHALMIC HERPES ZOSTER (Infections and infestations) | 0 | 0 | 0 | 1 | 0
ORAL CANDIDIASIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
ORCHITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
OTITIS MEDIA ACUTE (Infections and infestations) | 1 | 0 | 0 | 0 | 0
PARONYCHIA (Infections and infestations) | 0 | 0 | 0 | 1 | 0
PERINEAL ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
PHARYNGOTONSILLITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
PILONIDAL CYST (Infections and infestations) | 1 | 0 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 1 | 0 | 0 | 0 | 0
RELAPSING FEVER (Infections and infestations) | 0 | 0 | 0 | 1 | 0
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 1 | 0 | 0 | 0 | 0
SEPSIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
SIALOADENITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1
SINUSITIS BACTERIAL (Infections and infestations) | 0 | 0 | 0 | 1 | 0
SUPERINFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0
TAENIASIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1
TINEA PEDIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
TRICHOPHYTOSIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1
URETHRITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
VIRAL LABYRINTHITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
ASTHENIA (General disorders) | 19 | 9 | 4 | 23 | 4
DRUG INEFFECTIVE (General disorders) | 17 | 8 | 6 | 11 | 1
PYREXIA (General disorders) | 4 | 4 | 2 | 6 | 1
INFLUENZA LIKE ILLNESS (General disorders) | 9 | 2 | 1 | 2 | 2
THERAPEUTIC RESPONSE SHORTENED (General disorders) | 4 | 1 | 1 | 4 | 2
PAIN (General disorders) | 1 | 0 | 2 | 4 | 3
DRUG INTOLERANCE (General disorders) | 2 | 2 | 2 | 1 | 0
CHEST PAIN (General disorders) | 3 | 1 | 0 | 0 | 1
FATIGUE (General disorders) | 1 | 0 | 1 | 1 | 2
MALAISE (General disorders) | 1 | 1 | 1 | 0 | 1
CHILLS (General disorders) | 0 | 0 | 1 | 2 | 0
HYPERTHERMIA (General disorders) | 3 | 0 | 0 | 0 | 0
INFLAMMATION (General disorders) | 0 | 0 | 1 | 1 | 1
OEDEMA PERIPHERAL (General disorders) | 2 | 0 | 1 | 0 | 0
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 | 0 | 0 | 1 | 0
INJECTION SITE HYPERSENSITIVITY (General disorders) | 2 | 0 | 0 | 0 | 0
PERIPHERAL SWELLING (General disorders) | 1 | 0 | 0 | 1 | 0
THERAPEUTIC REACTION TIME DECREASED (General disorders) | 0 | 0 | 0 | 2 | 0
ADMINISTRATION SITE EXTRAVASATION (General disorders) | 1 | 0 | 0 | 0 | 0
ADVERSE DRUG REACTION (General disorders) | 0 | 1 | 0 | 0 | 0
ADVERSE EVENT (General disorders) | 0 | 0 | 0 | 1 | 0
CHEST DISCOMFORT (General disorders) | 1 | 0 | 0 | 0 | 0
CYST (General disorders) | 0 | 0 | 0 | 1 | 0
DISCOMFORT (General disorders) | 0 | 0 | 0 | 1 | 0
DISEASE PROGRESSION (General disorders) | 1 | 0 | 0 | 0 | 0
POLYP (General disorders) | 0 | 0 | 0 | 0 | 1
PUNCTURE SITE PAIN (General disorders) | 0 | 0 | 0 | 1 | 0
THERAPEUTIC RESPONSE DECREASED (General disorders) | 1 | 0 | 0 | 0 | 0
THERAPY NON-RESPONDER (General disorders) | 0 | 1 | 0 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 9 | 5 | 4 | 17 | 4
ABDOMINAL PAIN (Gastrointestinal disorders) | 12 | 4 | 1 | 6 | 2
VOMITING (Gastrointestinal disorders) | 9 | 3 | 2 | 2 | 2
CROHN'S DISEASE (Gastrointestinal disorders) | 10 | 0 | 0 | 1 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 6 | 2 | 0 | 3 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 | 0 | 1 | 4 | 1
NAUSEA (Gastrointestinal disorders) | 1 | 3 | 1 | 1 | 3
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 2 | 0 | 4 | 0
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 3 | 1 | 0 | 2 | 1
ODYNOPHAGIA (Gastrointestinal disorders) | 4 | 0 | 0 | 3 | 0
APHTHOUS ULCER (Gastrointestinal disorders) | 4 | 0 | 0 | 2 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 1
DYSPEPSIA (Gastrointestinal disorders) | 1 | 0 | 3 | 1 | 0
COLITIS ULCERATIVE (Gastrointestinal disorders) | 0 | 3 | 0 | 1 | 0
DRY MOUTH (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 2
TOOTHACHE (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 1
GASTROINTESTINAL MOTILITY DISORDER (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0
MUCOUS STOOLS (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0
SUBILEUS (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0
ANAL FISTULA (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
COLITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
DYSPHAGIA (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
ENTERITIS (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
GASTRITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
ILEAL STENOSIS (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
INTESTINAL ULCER (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
OESOPHAGITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
ABDOMINAL RIGIDITY (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
ANAL INCONTINENCE (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
ANORECTAL DISORDER (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
CHRONIC GASTRITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
COLITIS MICROSCOPIC (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
COLONIC FISTULA (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
DIARRHOEA HAEMORRHAGIC (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
DUODENITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
FAECES SOFT (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
FISTULA OF SMALL INTESTINE (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
FOOD POISONING (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
FREQUENT BOWEL MOVEMENTS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
GINGIVAL SWELLING (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
HIATUS HERNIA (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
ILEAL ULCER (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
INTRA-ABDOMINAL FLUID COLLECTION (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
PROCTALGIA (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
SMALL INTESTINAL STENOSIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
ULCERATIVE GASTRITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
PSORIASIS (Skin and subcutaneous tissue disorders) | 13 | 3 | 0 | 5 | 3
PRURITUS (Skin and subcutaneous tissue disorders) | 11 | 1 | 2 | 5 | 2
ECZEMA (Skin and subcutaneous tissue disorders) | 9 | 1 | 0 | 3 | 1
RASH (Skin and subcutaneous tissue disorders) | 6 | 2 | 2 | 0 | 1
SKIN LESION (Skin and subcutaneous tissue disorders) | 5 | 1 | 0 | 2 | 1
DRY SKIN (Skin and subcutaneous tissue disorders) | 7 | 0 | 0 | 0 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 4 | 2 | 0 | 2 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 3 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 1 | 0
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 0 | 1
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 0 | 1
ACNE (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 0
ERYTHROSIS (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
GUTTATE PSORIASIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
INTERTRIGO (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
MACULE (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
DERMAL CYST (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
DERMATITIS BULLOUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
DERMATITIS EXFOLIATIVE (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
DERMATOSIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
DIFFUSE ALOPECIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
ECZEMA WEEPING (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
ERYTHEMA NODOSUM (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
NAIL DYSTROPHY (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
NAIL PSORIASIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
ONYCHOLYSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
PAPULE (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
PITYRIASIS ROSEA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
PURPURA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
PUSTULAR PSORIASIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
ROSACEA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
SEBORRHOEIC DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
SKIN DEPIGMENTATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
SKIN HYPOPIGMENTATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 18 | 7 | 2 | 6 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 8 | 2 | 3 | 5 | 3
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0 | 3 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 4 | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 4 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 6 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 | 1
TENDON DISORDER (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 3 | 1
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0
LUPUS-LIKE SYNDROME (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0
TENDONITIS (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 0
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
SJOGREN'S SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
ANKYLOSING SPONDYLITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
CHONDROPATHY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
ENTHESOPATHY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
FISTULA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
INTERVERTEBRAL DISC DISORDER (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
LIMB DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
MENISCAL DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
RHEUMATIC DISORDER (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
SACROILIITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
SLIPPING RIB SYNDROME (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
SOFT TISSUE MASS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
SPINAL DISORDER (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
SPONDYLITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
SPONDYLOLYSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
TENOSYNOVITIS STENOSANS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
TRIGGER FINGER (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
HEADACHE (Nervous system disorders) | 18 | 6 | 4 | 9 | 4
PARAESTHESIA (Nervous system disorders) | 0 | 0 | 0 | 7 | 2
SCIATICA (Nervous system disorders) | 2 | 0 | 1 | 4 | 0
CERVICOBRACHIAL SYNDROME (Nervous system disorders) | 1 | 0 | 2 | 0 | 0
TREMOR (Nervous system disorders) | 2 | 0 | 0 | 1 | 0
CAROTID ARTERIOSCLEROSIS (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
HYPOAESTHESIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
MIGRAINE (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
PRESYNCOPE (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
SYNCOPE (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
AMNESIA (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
AURA (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
AXONAL NEUROPATHY (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
BURNING SENSATION (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
CEREBRAL ATROPHY (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
CERVICAL MYELOPATHY (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
CERVICAL RADICULOPATHY (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
COGNITIVE DISORDER (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
DROP ATTACKS (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
EPILEPSY (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
INTRACRANIAL ANEURYSM (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
NEURALGIA (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
OCCIPITAL NEURALGIA (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
PERIPHERAL SENSORIMOTOR NEUROPATHY (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
PETIT MAL EPILEPSY (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
SMALL FIBRE NEUROPATHY (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 4 | 12 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 1 | 3 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 2 | 0
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3 | 0
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
BRONCHIAL DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
BRONCHIAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
NASAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
TONSILLAR INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
VOCAL CORD INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 9 | 1 | 1 | 0 | 0
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 6 | 0
FALL (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 1 | 1
INJECTION RELATED REACTION (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0
EXPOSURE DURING BREAST FEEDING (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
LIMB INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
WOUND (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
ACCIDENT AT WORK (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
CARBON MONOXIDE POISONING (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
DRUG ADMINISTRATION ERROR (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
EPICONDYLITIS (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
EXPOSURE VIA FATHER (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
EYE BURNS (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
FOREIGN BODY IN EYE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
INAPPROPRIATE SCHEDULE OF DRUG ADMINISTRATION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
INTESTINAL ANASTOMOSIS COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
JOINT INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
MUSCLE RUPTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
NASAL INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
PROCEDURAL NAUSEA (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
SKIN WOUND (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
THERMAL BURN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
TOOTH AVULSION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
WOUND SECRETION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
WEIGHT DECREASED (Investigations) | 1 | 0 | 1 | 5 | 0
TRANSAMINASES INCREASED (Investigations) | 2 | 0 | 0 | 3 | 0
WEIGHT INCREASED (Investigations) | 4 | 0 | 0 | 0 | 1
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 | 1 | 2 | 1 | 0
DRUG SPECIFIC ANTIBODY PRESENT (Investigations) | 1 | 1 | 0 | 1 | 0
LIPIDS ABNORMAL (Investigations) | 0 | 0 | 0 | 3 | 0
EMERGENCY CARE EXAMINATION (Investigations) | 2 | 0 | 0 | 0 | 0
HEPATIC ENZYME INCREASED (Investigations) | 2 | 0 | 0 | 0 | 0
BONE SCAN ABNORMAL (Investigations) | 1 | 0 | 0 | 0 | 0
C-REACTIVE PROTEIN ABNORMAL (Investigations) | 0 | 0 | 1 | 0 | 0
C-REACTIVE PROTEIN INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0
CARDIAC MURMUR (Investigations) | 1 | 0 | 0 | 0 | 0
CARDIOVASCULAR EXAMINATION (Investigations) | 0 | 1 | 0 | 0 | 0
CREATININE RENAL CLEARANCE DECREASED (Investigations) | 0 | 0 | 1 | 0 | 0
ELECTROPHORESIS PROTEIN ABNORMAL (Investigations) | 0 | 0 | 0 | 0 | 1
GLOMERULAR FILTRATION RATE DECREASED (Investigations) | 0 | 0 | 1 | 0 | 0
HEPATIC ENZYME ABNORMAL (Investigations) | 1 | 0 | 0 | 0 | 0
SERUM FERRITIN DECREASED (Investigations) | 1 | 0 | 0 | 0 | 0
HEPATOCELLULAR INJURY (Hepatobiliary disorders) | 11 | 3 | 1 | 10 | 3
HEPATIC STEATOSIS (Hepatobiliary disorders) | 2 | 1 | 0 | 1 | 0
CHOLANGITIS SCLEROSING (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 0 | 0 | 0 | 2 | 0
CHOLESTASIS (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
HEPATITIS (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
HEPATOMEGALY (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
HYPERPLASTIC CHOLECYSTOPATHY (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
LIVER DISORDER (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
OPHTHALMIC HERPES ZOSTER (Eye disorders) | 0 | 0 | 0 | 1 | 0
DRY EYE (Eye disorders) | 3 | 0 | 1 | 0 | 1
CHALAZION (Eye disorders) | 0 | 0 | 1 | 2 | 1
UVEITIS (Eye disorders) | 1 | 1 | 0 | 2 | 0
CATARACT (Eye disorders) | 2 | 0 | 0 | 1 | 0
EYE PAIN (Eye disorders) | 2 | 0 | 0 | 1 | 0
CHORIORETINOPATHY (Eye disorders) | 0 | 0 | 0 | 2 | 0
OCULAR HYPERAEMIA (Eye disorders) | 1 | 0 | 0 | 1 | 0
ABNORMAL SENSATION IN EYE (Eye disorders) | 1 | 0 | 0 | 0 | 0
BLEPHARITIS (Eye disorders) | 1 | 0 | 0 | 0 | 0
CONJUNCTIVAL DISORDER (Eye disorders) | 0 | 0 | 0 | 1 | 0
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 0 | 1 | 0 | 0 | 0
EYE ALLERGY (Eye disorders) | 1 | 0 | 0 | 0 | 0
EYE IRRITATION (Eye disorders) | 1 | 0 | 0 | 0 | 0
EYE OEDEMA (Eye disorders) | 1 | 0 | 0 | 0 | 0
EYELID OEDEMA (Eye disorders) | 0 | 1 | 0 | 0 | 0
EYELID PTOSIS (Eye disorders) | 1 | 0 | 0 | 0 | 0
FOREIGN BODY SENSATION IN EYES (Eye disorders) | 1 | 0 | 0 | 0 | 0
KERATITIS (Eye disorders) | 1 | 0 | 0 | 0 | 0
LACRIMATION INCREASED (Eye disorders) | 1 | 0 | 0 | 0 | 0
VISION BLURRED (Eye disorders) | 1 | 0 | 0 | 0 | 0
RENAL COLIC (Renal and urinary disorders) | 6 | 1 | 0 | 4 | 1
DYSURIA (Renal and urinary disorders) | 1 | 1 | 0 | 5 | 0
POLLAKIURIA (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 1
CALCULUS URINARY (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
URINARY INCONTINENCE (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
BLADDER CYST (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
PELVI-URETERIC OBSTRUCTION (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
URINARY RETENTION (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
URINARY TRACT DISORDER (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
LYMPHOPENIA (Blood and lymphatic system disorders) | 4 | 2 | 0 | 1 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 3 | 1 | 1 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0 | 0
EOSINOPHILIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0
HYPERCOAGULATION (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
HYPERLEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
LYMPHADENITIS (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
URTICARIA CHRONIC (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
SOMNOLENCE (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 1 | 1 | 1 | 2 | 0
POLYURIA (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 2 | 1 | 0
IRON DEFICIENCY (Metabolism and nutrition disorders) | 8 | 1 | 0 | 0 | 0
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 4 | 0
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 3 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 0
GOUT (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
CELL DEATH (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
MULTI-VITAMIN DEFICIENCY (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
MOLE EXCISION (Surgical and medical procedures) | 1 | 0 | 1 | 1 | 0
ARTHRODESIS (Surgical and medical procedures) | 0 | 0 | 0 | 2 | 0
EVENTRATION REPAIR (Surgical and medical procedures) | 2 | 0 | 0 | 0 | 0
NASAL SEPTAL OPERATION (Surgical and medical procedures) | 0 | 2 | 0 | 0 | 0
ANGIOPLASTY (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
ARTIFICIAL CROWN PROCEDURE (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
BENIGN TUMOUR EXCISION (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
BUNION OPERATION (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
CAUTERY TO NOSE (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
CHOLECYSTECTOMY (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
DRAIN PLACEMENT (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
ENDODONTIC PROCEDURE (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
EYE LASER SURGERY (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
HAEMORRHOID OPERATION (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
HIP ARTHROPLASTY (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
ILEOCOLOSTOMY (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
ILEOSTOMY CLOSURE (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
KNEE ARTHROPLASTY (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
LAPAROTOMY (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
LIMB OPERATION (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
MENISCUS REMOVAL (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
PARONYCHIA DRAINAGE (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
PILONIDAL SINUS REPAIR (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
SKIN LESION EXCISION (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
STENT PLACEMENT (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
TURBINOPLASTY (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
URINARY INCONTINENCE SURGERY (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
VERTIGO (Ear and labyrinth disorders) | 6 | 1 | 1 | 8 | 1
EAR PAIN (Ear and labyrinth disorders) | 2 | 0 | 0 | 2 | 0
DEAFNESS BILATERAL (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
EXTERNAL EAR INFLAMMATION (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
HYPOACUSIS (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
OTORRHOEA (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
TYMPANIC MEMBRANE PERFORATION (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
DEPRESSION (Psychiatric disorders) | 4 | 0 | 0 | 1 | 0
INSOMNIA (Psychiatric disorders) | 4 | 0 | 0 | 0 | 0
ANXIETY DISORDER (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0
BURNOUT SYNDROME (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0
SLEEP DISORDER (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0
STRESS (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0
AFFECTIVE DISORDER (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
AGGRESSION (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
ANXIETY (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
BIPOLAR DISORDER (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
IRRITABILITY (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
PROSTATITIS (Reproductive system and breast disorders) | 0 | 0 | 0 | 4 | 0
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 | 1 | 0 | 0 | 0
CERVICAL DYSPLASIA (Reproductive system and breast disorders) | 2 | 0 | 0 | 0 | 0
METRORRHAGIA (Reproductive system and breast disorders) | 2 | 0 | 0 | 0 | 0
BREAST HAEMATOMA (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
BREAST PAIN (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
DYSPAREUNIA (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
ENDOMETRIOSIS (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
FIBROCYSTIC BREAST DISEASE (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
INFERTILITY (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
MENOMETRORRHAGIA (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
MENORRHAGIA (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
PELVIC PAIN (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
VULVAL ULCERATION (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
VULVOVAGINAL SWELLING (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
HYSTEROCELE (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
HYPERSENSITIVITY (Immune system disorders) | 2 | 2 | 0 | 4 | 1
DRUG HYPERSENSITIVITY (Immune system disorders) | 2 | 1 | 1 | 2 | 0
ANAPHYLACTIC REACTION (Immune system disorders) | 1 | 0 | 0 | 1 | 0
IMMUNODEFICIENCY (Immune system disorders) | 0 | 1 | 0 | 0 | 0
SEASONAL ALLERGY (Immune system disorders) | 0 | 1 | 0 | 0 | 0
TYPE IV HYPERSENSITIVITY REACTION (Immune system disorders) | 0 | 0 | 0 | 1 | 0
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 0 | 0 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 1 | 0 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 2 | 0
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0
CARCINOMA IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
SEBORRHOEIC KERATOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
HYPERTENSION (Vascular disorders) | 1 | 0 | 0 | 1 | 2
HOT FLUSH (Vascular disorders) | 2 | 0 | 0 | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 0 | 2 | 0
ARTERIOSCLEROSIS (Vascular disorders) | 0 | 0 | 0 | 1 | 0
HAEMATOMA (Vascular disorders) | 1 | 0 | 0 | 0 | 0
HYPOTENSION (Vascular disorders) | 1 | 0 | 0 | 0 | 0
PHLEBITIS (Vascular disorders) | 0 | 0 | 0 | 1 | 0
BRADYCARDIA (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
PALPITATIONS (Cardiac disorders) | 1 | 1 | 0 | 0 | 0
ANGINA PECTORIS (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
ARTERIOSPASM CORONARY (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
BUNDLE BRANCH BLOCK (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 2 | 1 | 0 | 1 | 0
BLIGHTED OVUM (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0
ECTOPIC PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0
GESTATIONAL DIABETES (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0
CORNEAL DYSTROPHY (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0
DERMOID CYST (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0
GILBERT'S SYNDROME (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0
PHIMOSIS (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0
HIRSUTISM (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
THYROID MASS (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
THYROIDITIS SUBACUTE (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
INVESTIGATION NONCOMPLIANCE (Social circumstances) | 0 | 0 | 0 | 1 | 0
TREATMENT NONCOMPLIANCE (Social circumstances) | 0 | 0 | 0 | 0 | 1
PRODUCT AVAILABILITY ISSUE (Product Issues) | 0 | 0 | 1 | 0 | 0
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
ABSCESS MANAGEMENT (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
ILEOSTOMY (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/38/NCT02925338/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/38/NCT02925338/SAP_001.pdf